CLINICAL TRIAL: NCT04767971
Title: Clinical Value of G-EYE Colonoscopy in Daily Practice for Adenoma Detection and Time for Polyp Removal
Status: Completed | Type: Observational
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Ralf Kiesslich, Prof., Dr. Horst Schmidt Klinik GmbH
Other Study IDs: G-EYE
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Adenoma; Colo-rectal Cancer
Keywords: Adenoma; Colorectal Cancer
MeSH Terms: conditions — Adenoma; Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Colonoscopy: Colonoscopy with a standard colonoscope
  Interventions: Device: Standard Colonoscopy
- G-EYE® Colonoscopy: Colonoscopy with a G-EYE Colonoscopy
  Interventions: Device: G-EYE Colonoscopy

INTERVENTIONS:
Device: Standard Colonoscopy — Colonoscopy with a standard colonoscope
  Groups: Standard Colonoscopy
Device: G-EYE Colonoscopy — Colonoscopy with a G-EYE Colonoscope
  Groups: G-EYE® Colonoscopy

SUMMARY:
Colonoscopy parameters will be compared before the introduction of the G-EYE endoscope and after the introduction of the G-EYE endoscope

DETAILED DESCRIPTION:
Colonoscopy parameters such as demographics, findings and procedural times will be compared before the introduction of the G-EYE endoscope and after the introduction of the G-EYE endoscope

ELIGIBILITY:
Inclusion Criteria:

- Indication for screening or surveillance colonoscopy based on the German guideline for colon cancer screening

Exclusion Criteria:

* Emergency procedure
* Patients with known inflammatory bowel diseases
* Patients with hereditary cancer syndromes
* Patients with acute colonic inflammation (e.g. diverticulitis, ischemic colitis)
* Patients after radiation of the abdomen or pelvis
* Patients with colonic surgery (except appendectomy)
* Patients with incomplete colonoscopy
* Patients with insufficient bowel preparation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Screening and surveillance colonoscopy patients
Sampling Method: Probability Sample
Enrollment: 2795 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Detection rate - measured by adenoma detection rate (% subjects having at least 1 adenoma) | February 2021
  G-EYE® colonoscopy adenoma detection rate compared to adenoma detection rate of standard colonoscopy
Effectiveness of intervention - measured by polyp removal time (mm:ss) | February 2021
  G-EYE® colonoscopy polyp removal time compared to polyp removal time of standard colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken Wiesbaden
Locations (1):
- Helios Dr. Horst Schmidt Kliniken, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: No